CLINICAL TRIAL: NCT00499499
Title: A Phase I Open-Label, Single-Arm, Dose Escalation Study of E7107 Administered Intravenously on Days 1 and 8 Every 21 Days to Patients With Solid Tumors
Brief Title: A Dose Escalation Study of E7107 Administered Intravenously on Days 1 and 8 Every 21 Days to Patients With Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Daniel Rossignol, Ph.D, Eisai Medical Research Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7107-A001-101
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Cancer
Keywords: Cancer; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — E 7107

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7107

INTERVENTIONS:
Drug: E7107 — E7107 will be administered as an intravenous infusion over 30 minutes at a starting dose of 0.6 mg/m^2 to the first cohort of patients. The same dose will be given on Days 1 and 8 of a 21-day cycle. Dose escalation will not occur until the maximum tolerated dose is reached. The selection of subsequent dose levels will be performed according to an accelerated design.

SUMMARY:
The purpose of this study is to investigate E7107 in patients with solid tumors. This is an open label, dose-escalation study of E7107. The maximum tolerated dose (MTD) of the single agent will be established by determining the occurrence of dose limiting toxicities during the first three weeks of therapy (Cycle 1). Patients in this study will be treated at multiple dose levels, starting at 0.6 mg/m^2. Patients will receive E7107 as a 30-minute intravenous infusion on Days 1 and 8 every 21 Days.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all of the inclusion criteria outlined below in order to be eligible to participate in the study.

1. Patients with histologically and/or cytologically confirmed solid tumors who have progressed after receiving approved therapies for their disease and for whom no effective therapies are available.
2. Surgery and radiotherapy must have been completed at least four weeks prior to study entry, and prior chemotherapy and other anti-cancer therapy, excluding bisphosphonates at a steady dose level, must have been discontinued 2 to 3 weeks previously. All acute toxicities related to these treatments must have resolved.
3. Aged ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. Written informed consent prior to any study specific screening procedures, which will include mandatory consent to provide a blood sample specifically for pharmacogenomic analysis, with the understanding that the patient may withdraw consent at any time without prejudice. Tumor biopsy for pharmacogenomic (PG) analysis will be voluntary.
6. Willing and able to comply with the protocol for the duration of the study.
7. Anticipated life expectancy > three months.

EXCLUSION CRITERIA:

Patients with the following characteristics will not be eligible for the study.

1. Symptomatic or progressive brain tumors or brain or leptomeningeal (CNS) metastases requiring clinical intervention, except if they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least two weeks before starting treatment with E7107.
2. Any of the following laboratory parameters:

   1. hemoglobin < 9 g/dL (5.6 mM)
   2. neutrophils < 1.5 x 10^9/L
   3. platelets < 100 x 10^9/L
   4. serum bilirubin > 25 μM (1.5 mg/dL)
   5. liver function tests (defined as AST and ALT) with values > 3 x ULN (5 x ULN if liver metastases are present)
   6. serum creatinine > 1.5 x ULN or creatinine clearance < 40 mL/min.
3. Positive history of HIV, active hepatitis B or active hepatitis C or severe/uncontrolled intercurrent illness or infection.
4. Clinically significant cardiac impairment or unstable ischemic heart disease (greater than Class II according to New York Heart Association (NYHA) classification) including a myocardial infarction within six months of study start.
5. Bleeding or thrombotic disorders, or using therapeutic dosages of anticoagulants
6. History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the Investigator, would impair study compliance.
7. Women who are pregnant or breast-feeding. Women of childbearing potential with either a positive serum pregnancy test at screening, a positive urine pregnancy test at the beginning of any cycle, or no pregnancy test. Women of childbearing potential unless using two forms of contraception, one of which must be a barrier method. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
8. Fertile men and fertile women who are not willing to use contraception, or fertile men or fertile women with a partner who is not willing to use contraception
9. Patients with a marked screening or baseline prolongation of QT/QTc interval using the Fridericia formula (ie, repeated demonstration of a QTc interval > 450 msec); a history of additional risk factors for Torsade de Pointe (e.g., heart failure, hypokalaemia, history of Long QT Syndrome).
10. Patients who have had radiation to >= 25% of their bone marrow (e.g., pelvic radiation).
11. Patients who have a history of previous Grade 2 or higher hypersensitivity to pladienolide B or derivatives and excipients of the formulation
12. Patients with significant comorbid disease or condition, which in the Investigator's opinion would exclude the patient from the study
13. Patients who have received an organ allograft ie, requiring immunosuppressive therapy
14. Beginning two weeks prior to dosing, patients are not allowed to take drugs that are strong CYP inhibitors (including grapefruit juice and herbal supplements) or inducers (including herbal supplements), or are metabolized by cytochrome P (CYPs) and known to have a narrow therapeutic window.
15. After MTD has been reached: Second malignancy within the past 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Tumor assessments should be performed at screening and then every 2 cycles. A best response according to RECIST (Response Evaluation Criteria in Solid Tumors) will be documented by the investigator for each patient. | Every 6 weeks

SECONDARY OUTCOMES:
Clinical examination (either full or symptom-directed), adverse event reporting, laboratory screens, and electrocardiograms (ECGs) will be performed at every visit. | Every 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Matczak, Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - Karmanos Cancer Center, Detroit, Michigan
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hong DS, Kurzrock R, Naing A, Wheler JJ, Falchook GS, Schiffman JS, Faulkner N, Pilat MJ, O'Brien J, LoRusso P. A phase I, open-label, single-arm, dose-escalation study of E7107, a precursor messenger ribonucleic acid (pre-mRNA) splicesome inhibitor administered intravenously on days 1 and 8 every 21 days to patients with solid tumors. Invest New Drugs. 2014 Jun;32(3):436-44. doi: 10.1007/s10637-013-0046-5. Epub 2013 Nov 22. PMID 24258465